CLINICAL TRIAL: NCT06957028
Title: CGM for the Early Detection and Management of Hyperglycemia in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); DexCom, Inc. (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IMAGINE
Record Dates: First submitted 2025-04-02; First posted 2025-05-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: GDM; CGM; Pregnancy
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Masking Description: Participants are initially masked from glucose results from continuous glucose monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose Lowering Group (Experimental)
  Interventions: Other: Diabetes Treatment
- Usual Care Group (with periodic blinded CGM) (Active Comparator)
  Interventions: Other: Usual Care Group
- Observational (No Intervention)

INTERVENTIONS:
Other: Diabetes Treatment — Management will include an unblinded CGM sensor worn 24/7, GDM specific nutrition information, training on using CGM in daily glucose management to achieve euglycemia (maximizing time 63-140 mg/dL [3.5-7.8 mmol/L]).
  Visits (which could be telehealth) per usual obstetrical care for glycemia management (expected to be about every 4 weeks for most participants) and weekly glycemic management with review of CGM data by site and by central CGM Resource Center for flagged cases.
  Participants not receiving glucose lowering medication by 24-28 weeks will undergo OGTT per usual obstetrical management and those with positive OGTT will be treated for GDM per usual clinic routine and continue to wear an unblinded CGM.
  Other Names: Continuous Glucose Monitoring
  Arms: Glucose Lowering Group
Other: Usual Care Group — The control group will receive usual obstetrical care at the clinical center. A general pregnancy nutrition information handout will be provided to each participant and a blinded CGM sensor will be placed at routine obstetrical care visits and worn for 10-14 days each time throughout the pregnancy beginning between 18-22 weeks' gestation.
  At 18-22 weeks, blinded CGM data will be reviewed to assess if participant has ≥25% time >140 mg/dL to determine if an early OGTT or glycemic management is required. Site clinicians will be unblinded to the masked CGM data for participants with CGM data ≥25% time >140 mg/dL and those participants may be treated as those with a positive OGTT.
  An OGTT will be performed at ~24-28 weeks per the clinic's usual routine and those with positive OGTT will be treated for GDM per usual clinic routine. If real-time CGM is to be used, then unblinded study CGM sensors can be used instead of blinded sensors for the duration of the study.
  Other Names: Blinded Continuous Glucose Monitoring
  Arms: Usual Care Group (with periodic blinded CGM)

SUMMARY:
The goal of this clinical trial is to use continuous glucose monitoring (CGM) to quickly detect and manage high blood sugar in pregnant women, early in pregnancy. The main questions it aims to answer are:

(1) any problems for the baby, such as being too large for their age, shoulder injuries (like broken bones), high bilirubin levels needing light treatment, low blood sugar, or needing to stay in the NICU; (2) any high blood pressure issues for the mother during pregnancy.

DETAILED DESCRIPTION:
Data from continuous glucose monitoring (CGM) in the Glucose Lowering group tracked over time, will be compared to data from blinded sensors in the Usual Care group approximately every 4 weeks.

* Pregnant women who do not have diabetes and have a single, uncomplicated pregnancy will be enrolled by 14 weeks and 6 days. They will start by wearing a hidden CGM sensor to check for high blood sugar.
* The blinded CGM sensor data will be evaluated to determine if the following criterion is met: 5% to <25% of values >140 mg/dL

  • An initial assessment will be made after 5 days and for those not meeting the criterion, again after 10 days
* Participants meeting the CGM hyperglycemia criteria and the other study eligibility criteria will proceed to randomization, which must be performed by 16 weeks 6 days of gestation.
* Participants who do not meet the CGM hyperglycemia criteria will form an observational cohort, provided that HbA1c is <6.5% (48 mmol/mol)

ELIGIBILITY:
Inclusion Criteria

1. Maternal age of 18 years and older
2. Singleton pregnancy
3. Gestational age up to 14w 6d of pregnancy, determined on ultrasound, for initiation of screening

   • Although it is preferable that ultrasound results be available prior to enrollment, if ultrasound results are not available at the time of enrollment, participant can have CGM initiated but will be dropped if not eligible after results are available
4. HbA1c <6.5% (48 mmol/mol) since onset of pregnancy

   • If HbA1c result not available at time of enrollment, participant can have blinded screening CGM initiated, but results will be needed prior to randomization to verify eligibility.
5. No prior history of gestational diabetes mellitus (GDM)
6. Able to read English or Spanish

Exclusion Criteria

1. Signs of abnormal fetal or placental development (suspected fetal anomaly or placenta accreta spectrum, low PAPPA) at first routine prenatal visit/ultrasound
2. Planned termination of pregnancy or any indications of miscarriage
3. Prior gastric bypass surgery
4. Pregravid diabetes (type 1 or type 2)
5. Unwillingness/inability to wear CGM sensor
6. Unwillingness to attend routine antenatal obstetric appointments
7. Use of corticosteroids by a route that can produce hyperglycemia (e.g., oral, intravenous, intramuscular, intra-articular) during the 7 days prior to initiating CGM screening or during the CGM screening

   • Topical and inhaled corticosteroids are acceptable
8. Use of insulin during the pregnancy prior to enrollment
9. Use of metformin within one week of the initiation of the blinded CGM sensor for screening or use of a GLP-1 or other weight-reduction medication that can affect glucose levels within 4 weeks of the initiation of the blinded CGM sensor for screening
10. Deemed unable to participate for medical reasons identified by their physician

Additional Criteria for RCT Eligibility

1. Screening CGM meeting study criteria for hyperglycemia: 5% to <25% time >140 mg/dL
2. Randomization by 16 week 6 days of pregnancy
3. No participation in a separate intervention trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of child bearing potential
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-11-27 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint of Neonatal Complications or Maternal Hypertensive Disorder of Pregnancy | Baseline to 45 weeks
  Composite endpoint of (1) neonatal complications of large for gestational age (LGA), shoulder dystocia (including humeral or clavicular fracture), elevated bilirubin requiring phototherapy, or neonatal intensive care unit (NICU) admission; or (2) maternal hypertensive disorder of pregnancy (HDP) .

SECONDARY OUTCOMES:
Composite of Neonatal Complications, Death, and Maternal Complications | Baseline to 45 weeks
  * Composite of neonatal complications
  * Individual maternal and neonatal complications
  * Neonatal death

OTHER OUTCOMES:
Small for Gestational Age Birth Weight | Baseline to 45 weeks
  Small for gestational age birth weight (<10th percentile)
CGM-Measured Time Less Than 54 mg/dL | Through study completion, an average of 30 months
  CGM-measured time less than 54 mg/dL (during comparative periods where Usual Care group has blinded CGM)
Severe Hypoglycemia Events | Through study completion, an average of 30 months
  Severe Hypoglycemia Events

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Durnwald, MD, Study Chair — University of Pennsylvania
Locations (10):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Emory University, Decatur, Georgia
  - IDC at Park Nicollet, Saint Louis Park, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds, Leeds
  - Norfolk and Norwich University Hospitals NHS, Norwich, Norwich

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT06957028/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT06957028/SAP_001.pdf
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT06957028/ICF_002.pdf